CLINICAL TRIAL: NCT01420211
Title: Influence of the OATP1B1 and OATP1B3 Genotype on the Hepatic Uptake of Primovist® in Healthy Volunteers and in Patients With Liver Disease
Brief Title: Influence of the OATP1B1 and OATP1B3 Genotype on the Hepatic Uptake of Primovist®
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Prof. Dr. W. Siegmund, MD, Clinical Pharmacology at the University of Greifswald
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Primovist - OATP1B1
Record Dates: First submitted 2011-08-16; First posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Pharmacokinetics; MRI; Liver; Drug Transporter; Gd-EOB-DTPA
Keywords: pharmacokinetics; MRI; liver; drug transporter; Gd-EOB-DTPA
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primovist (Experimental)
  Interventions: Drug: Primovist® 0,25 mmol/ml solution for injection; Device: MRI

INTERVENTIONS:
Drug: Primovist® 0,25 mmol/ml solution for injection — intravenous bolus injection of 25 µmol/kg (=0,1 ml/kg) body weight Primovist® and blood sampling before (serum blank) and 6, 11, 21, 31, 45, 65, 95, 125 min and 3, 4, 6, 8, 12, 24 and 48 h after drug administration
Device: MRI — lmaging of 20 slices (thickness: 3 mm; max. time of imaging 10 s) before and 0.25, 1, 2, 3, 4, 5, 7, 8, 9, 10, 20, 30, 40, 50, 60, 90 and 120 min after intravenous bolus injection of 25 µmol/kg (=0,1 ml/kg) body weight Primovist®

SUMMARY:
The objective of the study is to assess the hepatic uptake of Primovist® after intravenous administration of 25 µmol/kg body weight in 56 healthy volunteers and in 60 patients with a liver disease in dependence on the OATP1B1- and OATP1B3-genotype.

DETAILED DESCRIPTION:
Gadolinium-ethoxybenzyl-diethylenetriamine-pentaacetic acid (Gadoxetate, Gd-EOB-DTPA, Primovist®) is a newly developed paramagnetic hepatobiliary contrast agent for magnetic resonance imaging (MRI) based on the extracellular fluid marker gadopentetate (Magnevist®). After intravenous administration, Gd-EOB-DTPA distributes rapidly within the intravascular and extracellular spaces and is taken up selectively by hepatocytes. The compound is eliminated from the blood and from the body mainly by two pathways: glomerular filtration of the kidneys and hepatobiliary excretion. There is many evidence that the hepatic uptake of Gd-EOB-DTPA from the sinusoidal blood is influenced by specific hepatic transporters of the organic anion transporter (OATP) family.

For the highly liver specific agent has been demonstrated that it markedly improves the quality of detection of focal liver lesions (adenoma, focal nodular hyperplasia, hepatocellular carcinoma). Because gadoxetate is taken up both in the normal liver parenchyma as well as in focal liver lesions of hepatocellular origin, it allows to distinguish between hepatocyte-containing and non-hepatocyte-containing tissue. In some indications (e.g. preoperative evaluation of patients with hepatocellular carcinoma), liver-specific contrast media like Gd-EOB-DTPA are superior to biphasic spiral computertomography.

Hepatic enhancement after intravenous administration of Gd-EOB-DTPA is known to be inhibited by bromosulfophthalein, taurocholate and rifampicin. Obviously, Gd-EOB-DTPA and other drugs compete for the organic anion transporters of the hepatocytes. In Oatp1 cRNA injected oocytes of Xenopus leavis, a saturable uptake of gadoxetic acid has been demonstrated. Since the human organic anion transporting polypeptide (OATP) 1B1 (previous names: OATP-C, L-ST1, OATP2), which is responsible for the hepatic uptake of several endogenous and exogenous compounds like bile acids, bilirubin, peptides, steroid conjugates, thyroid hormones, methotrexate, statins and ezetimibe, is predominantly expressed in the basolateral membrane of hepatocytes, Gd-EOB-DTPA might be a substrate of this uptake transporter.

Because there were described functional relevant single nucleotide polymorphisms (SNP) for OATP1B1, which were responsible for markedly reduced transporter function and which were even shown to alter plasma concentrations of pravastatin and ezetimibe in vivo, we want to investigate the impact of several genotypes of OATP1B1 on disposition of Gd-EOB-DTPA. While *15 and *5 carriers of OATP1B1 were described to exhibit decreased lipid-lowering potency and increased statin-induced myopathy, *1b carriers exerted a significantly reduced bioavailability of ezetimibe. Due to the fact that the interesting haplotypes like OATP1B1 *15 and *1b are in fact relatively common in European subjects, we intend to define its influence on Gd-EOB-DTPA pharmacokinetics and on different signal intensities in magnetic resonance imaging of the liver.

OATP 1B3 (previous names: OATP8,LST-2), which is also predominantly expressed in the basolateral membrane of hepatocytes, is responsible for the hepatic uptake of several endogenous and exogenous compounds like bile acids, 17β-glucuronosyl estradiol, BSP or digoxin.

There is evidence from very recent experimental studies in our laboratory, that Primovist® is not only a substrate of OATP1B1 but also of the second liver specific uptake transporter OATP1B3. The MRT contrast agent inhibits the uptake of BSP in HEK tansfected with human OATP1B1 and OATP1B3 and it is also better taken up by these cells than by non-transfected parental cells. Therefore, we concluded that OATP1B3 might be additionally to OATP1B1 an specific uptake transporter in human liver.

Very recently, at least six single nucleotide polymorphisms (SNP) of OATP1B3 have been described in literature. At least two of them were described to be of functional relevance: 334T>G (Ser112Ala) and 699G>A (met233Ile). The allele frequencies of the 334T>G and 699G>A variants in European Caucasians were reported to be 74 % and 71%, respectively.

The influence of these amino-acid substitutions on OATP1B3 transport function and cellular localization seems to be substrate and cell line dependent. In man, it was shown that OATP1B3*2 influences obviously the hepatic uptake of erythromycin and hence the results of the ERMBT (erythromycin breath test) in cancer patients.

Therefore, carriers of OATP1B3 334T>G and OATP1B3 699G>A are planned to be included into the study with Primovist® to confirm whether the selective hepatic uptake carrier OATP1B3 is involved in hepatic uptake of the MRI contrast agent additionally to OATP1B1.

In several animal studies a reduced enhancement of Gd-EOB-DTPA was observed in acute hepatitis, fatty liver and cholestasis models. Obviously the hepatic uptake of gadexotate might be determined by liver diseases which lead to an altered function of hepatocytes. Therefore it is a further aim of the study to assess the influence of liver diseases on Gd-EOB-DTPA pharmacokinetics and signal intensity and its possible modification by the OATP1B1-genotype in 60 patients which are subjected to MR imaging of the liver.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years
* sex: male and female
* ethnic origin: white
* body weight: 19 to 27 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent

Exclusion Criteria:

* weight less than 45 kg
* claustrophobia
* cardiac pacemakers, metallic implants or metal-containing tatoos
* history of allergic reactions, allergic deseases (e.g. asthma bronchiale)
* known hypersensitivity to the study medication or to their adjuvants
* existing cardiac or hematological diseases and/or pathological findings, which might interfere with the drug's safety, tolerability and/or pharmacokinetics
* existing hepatic and renal diseases and/or pathological findings, which might interfere with the drug's safety, tolerability and/or pharmacokinetics
* existing gastrointestinal diseases and/or pathological findings, which might interfere with the drug's safety, tolerability and/or pharmacokinetics
* acute or chronic diseases which could affect drug metabolism or elimination
* history of any serious psychological disorder
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* positive anti-HIV-test, HBs-Ag-test or anti-HCV-test
* volunteers who are on a diet which could affect the pharmacokinetics of the drug
* heavy tea or coffee drinkers (more than 1L per day)
* lactation and pregnancy test positive or not performed
* volunteers suspected or known not to follow instructions
* volunteers who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* volunteers liable to orthostatic dysregulation, fainting, or blackouts
* participation in a clinical trial during the last 3 months prior to the start of the study
* less than 14 days after last acute disease
* any systemically available medication within 4 weeks prior to the intended first administration unless because of the terminal elimination half-life complete elimination from the body can be assumed for the drug and/or its primary metabolites (except oral contraceptives)
* repeated use of drugs during the last 4 weeks prior to the intended first administration, which can influence hepatic biotransformation (e.g. barbiturates, cimetidine, phenytoin, rifampicin)
* intake of grapefruit containing food or beverages within 7 days prior to administration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2006-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic characteristics | before (serum blank) and 6, 11, 21, 31, 45, 65, 95, 125 min and 3, 4, 6, 8, 12, 24 and 48 h after drug administration
  AUC0-t is calculated by the trapezoidal formula. AUC0-t is assessed up to the last sampling time above the limit of quantitation and is extrapolated to infinity using standard techniques. Cmax and Tmax will be obtained directly from the measured concentration-time curves. t1/2 will be evaluated from the terminal slope by log-linear regression analysis.
signal intensity of liver | before and 0.25, 1, 2, 3, 4, 5, 7, 8, 9, 10, 20, 30, 40, 50, 60, 90 and 120 min after drug administration
  Dynamic enhanced MR examination with 0.1ml/kg/KG (flow:2ml/s) Gd-EOB-DTPA and breath-hold gradient-echo T1-weighted VIBE images (Volumen interpolated breathhold examination) will be acquired on the 1.5T MRI (Siemens Symphony maestro class). Time of imaging can be seen on the time schedule. The SNR and the time to maximum enhancement will be calculated for each organ.

SECONDARY OUTCOMES:
signal intensity of gallbladder | before and 0.25, 1, 2, 3, 4, 5, 7, 8, 9, 10, 20, 30, 40, 50, 60, 90 and 120 min after drug administration
  Dynamic enhanced MR examination with 0.1ml/kg/KG (flow:2ml/s) Gd-EOB-DTPA and breath-hold gradient-echo T1-weighted VIBE images (Volumen interpolated breathhold examination) will be acquired on the 1.5T MRI (Siemens Symphony maestro class). Time of imaging can be seen on the time schedule. The SNR and the time to maximum enhancement will be calculated for each organ.
signal intensity of background noise | before and 0.25, 1, 2, 3, 4, 5, 7, 8, 9, 10, 20, 30, 40, 50, 60, 90 and 120 min after drug administration
  Dynamic enhanced MR examination with 0.1ml/kg/KG (flow:2ml/s) Gd-EOB-DTPA and breath-hold gradient-echo T1-weighted VIBE images (Volumen interpolated breathhold examination) will be acquired on the 1.5T MRI (Siemens Symphony maestro class). Time of imaging can be seen on the time schedule. The SNR and the time to maximum enhancement will be calculated for each organ.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology at the University of Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany